CLINICAL TRIAL: NCT04527575
Title: Simple, Blind, Placebo-controlled, Randomized Study of the Safety, Reactogenicity and Immunogenicity of Vaccine Based on Peptide Antigens for the Prevention of COVID-19 (EpiVacCorona), in Volunteers Aged 18-60 Years (I-II Phase)
Brief Title: Study of the Safety, Reactogenicity and Immunogenicity of "EpiVacCorona" Vaccine for the Prevention of COVID-19
Acronym: EpiVacCorona
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Federal Budgetary Research Institution State Research Center of Virology and Biotechnology "Vector" (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: COV/pept-01/20
Record Dates: First submitted 2020-08-11; First posted 2020-08-26 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Covid19
Keywords: Covid19; SARS-CoV-2; EpiVacCorona; vaccination
MeSH Terms: conditions — COVID-19 | interventions — EpiVacCorona vaccine; Solvents

STUDY DESIGN:
Intervention Model Description: Simple, blind, placebo-controlled, randomized study involving healthy volunteers
Who Masked: Participant, Investigator
Masking Description: Masking in Phase 2
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- "EpiVacCorona" (An Open Study) (Experimental): Group 1: 14 volunteers who will be vaccinated with the EpiVacCorona vaccine twice spaced 21 days apart, intramuscularly, at a dose of 0.5 ml
  Interventions: Biological: EpiVacCorona (EpiVacCorona vaccine based on peptide antigens for the prevention of COVID-19)
- "EpiVacCorona" (A Simple, Blind, Randomized Study) (Experimental): Group 2: Administration of the EpiVacCorona vaccine, intramuscularly, twice, 21 days spaced apart, at a dose of 0.5 ml (43 volunteers)
  Interventions: Biological: EpiVacCorona (EpiVacCorona vaccine based on peptide antigens for the prevention of COVID-19)
- "Placebo" (A Simple, Blind, Randomized Study) (Placebo Comparator): Group 3: Тhe use of placebo (sodium chloride, solvent for the preparation of dosage forms for injection 0.9%) intramuscularly twice space 21 days apart at a dose of 0.5 ml (43 volunteers)
  Interventions: Other: Placebo (sodium chloride bufus, solvent for the preparation of dosage forms for injection 0.9%)

INTERVENTIONS:
Biological: EpiVacCorona (EpiVacCorona vaccine based on peptide antigens for the prevention of COVID-19) — EpiVacCorona vaccine is intended to prevent COVID-19. The vaccine relies on chemically synthesized peptide antigens of SARS-CoV-2 proteins, conjugated to a carrier protein and adsorbed on an aluminum-containing adjuvant (aluminum hydroxide). The EpiVacCorona vaccine contributes to the development of protective immunity against SARS-CoV-2 coronavirus following two intramuscular administrations spaced 21-28 days apart.
  Arms: "EpiVacCorona" (A Simple, Blind, Randomized Study); "EpiVacCorona" (An Open Study)
Other: Placebo (sodium chloride bufus, solvent for the preparation of dosage forms for injection 0.9%) — The use of placebo: intramuscularly, twice, spaced 21 days apart, at a dose of 0.5 ml (43 volunteers)
  Arms: "Placebo" (A Simple, Blind, Randomized Study)

SUMMARY:
The aim of the clinical study is to determine the safety, reactogenicity and immunogenicity parameters of the EpiVacCorona vaccine in volunteers aged 18-60 years.

The research tasks are to:

* evaluate the safety of the EpiVacCorona vaccine when administered twice intramuscularly;
* evaluate the reactogenicity of the EpiVacCorona vaccine when administered twice intramuscularly;
* identify the development of adverse reactions to vaccine administration;
* study the humoral and cellular immune responses following two doses of the EpiVacCorona vaccine.

DETAILED DESCRIPTION:
The first phase of the clinical trial is an open trial. The study will enroll 14 men and women aged 18 to 30 years, inclusive, who meet the inclusion criteria and have no exclusion criteria, whose data will be used for subsequent analysis of safety and immunogenicity.

The second phase of the clinical trial is a simple, blind, placebo-controlled, randomized, parallel-group study. The study will enroll 86 men and women aged 18 to 60 years, inclusive, who meet the inclusion criteria and have no exclusion criteria whose, the data will be used for subsequent analysis of safety and immunogenicity.

If volunteers drop out of the study, they will not be replaced.

ELIGIBILITY:
1. Availability of a signed and dated informed consent of the volunteer to participate in a clinical trial, prior to any of the study procedures.
2. Verified diagnosis is "healthy" according to the data of the standard clinical, laboratory and instrumental examination methods.
3. Age from 18 to 60 years old inclusive.
4. Body mass index from 18.5 to 30 kg / m3.
5. Ability to attend all scheduled visits and all planned procedures and examinations.
6. Consent of volunteers to use effective contraceptive methods throughout the study, including the observation period for possible post-vaccination reactions.

Exclusion Criteria:

1. Contacts with COVID-19 patients for 14 days prior to the start of the clinical trial.
2. Hypersensitivity to any component of the product, allergy to the components of the vaccine.
3. The history of allergic reactions to any vaccination in the past.
4. Serious post-vaccination reactions/complications associated with any vaccination in the past.
5. Pregnancy and breastfeeding.
6. Military personnel on conscription.
7. Persons detained in pre-trial detention facilities and those serving sentences in prison.
8. Children under the age of 18.
9. Symptoms of any disease at the time of inclusion in the study or if it has passed less than 4 weeks since recovery.
10. The history of any acute respiratory disease within less than 3 months prior to inclusion in the study.
11. The history of acute infectious or non-communicable diseases, exacerbation of chronic diseases within less than 4 weeks before the start of the study.
12. The history of tuberculosis (pulmonary and extrapulmonary), cancer, autoimmune diseases, skin diseases (pemphigus, psoriasis, eczema, atopic dermatitis).
13. Long-term use (more than 14 days) of immunosuppressive drug, systemic glucocorticosteroids or immunomodulatory drugs within 6 months prior to the study.
14. Vaccination with any vaccine within one month prior to vaccination.
15. Taking immunoglobulin drugs or blood products within last 3 months prior to the study.
16. The history of treatment with human immunoglobulin drugs within, less than 6 months since such treatment.
17. Donation (450 ml of blood or plasma and more) within less than 2 months prior to the study.
18. Acute or chronic diseases of the cardiovascular, bronchopulmonary, neuroendocrine system, as well as diseases of the gastrointestinal tract, liver, kidneys, surgery on the gastrointestinal tract (except appendectomy).
19. The history of participation in other clinical trials within less than 3 months prior to the start of this study.
20. Individuals with alcohol, drug dependence or drug addiction. Taking more than 10 units of alcohol per week (1 unit of alcohol is equivalent to 1/2 litre of beer, 200 ml of wine or 50 ml of alcohol) or anamnestic information about alcoholism, drug addiction, and substance misuse. Individuals with positive results of urine examination for drugs and/or with alcohol findings in the exhaled air during the visits.
21. Mental illness and neurasthenia.
22. Non-compliance with the inclusion criteria.
23. Women in the premenopausal period (the last menstruation ≤ 1 year prior to the signing of informed consent) who are not surgically sterile and women who have reproductive potential, but do not use acceptable birth controls or do not plan to use them throughout the study and do not agree to a urine test for pregnancy during the participation in the study.
24. Positive test for HIV, viral hepatitis B and C, lues venerea.
25. Other comorbidities that the researcher believes may interfere with the evaluation of the study's objectives.

And:

1. The researcher's decision to exclude the volunteer for the benefit of the volunteer.
2. False inclusion (violation of inclusion and non-inclusion criteria) or the appearance of non-inclusion criteria during the study.
3. The decision of the researcher or the Customer to exclude the volunteer from the study due to a clinically significant deviation from the protocol/violation of the protocol.
4. Any undesirable phenomenon requiring the appointment of drugs not authorized by the protocol of this study.
5. Refusal of a volunteer to continue to participate in the study or his/her indiscipline.
6. Volunteer's desire to complete the study early for any reason.
7. Volunteer's failure to show up for a scheduled visit without the researcher's warning or loss of communication with the volunteer.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
The proportion of vaccinated volunteers with no laboratory confirmed symptoms caused by SARS-CoV-2 within 9 months post vaccination | throughout the study, an average of 270 days
  • The proportion of vaccinated volunteers with no laboratory confirmed symptoms caused by SARS-CoV-2, in combination with one or more of the following symptoms: fever or chills; cough; shortness of breath or labored breathing; fatigue; muscle pain; headache; The proportion of vaccinated volunteers with no laboratory confirmed symptoms caused loss of taste or smell; sore throat; a stuffy nose or runny nose; nausea or vomiting; diarrhea, within 9 months post vaccination versus a placebo.

SECONDARY OUTCOMES:
The proportion of volunteers with increased levels of the immune response in terms of geometric mean titers of specific antibodies in ELISA following the vaccination compared with a placebo. | at days 0, 1, 14, 20, 35, 42, 90, 180, 270
  • The proportion of volunteers with increased levels of the immune response in terms of geometric mean titers of specific antibodies in ELISA greater ≥ 4 times 21 days following the second vaccination and 90, 180 and 270 days following the first vaccination compared with a placebo.
The proportion of volunteers with increased levels of the immune response in terms of specific neutralizing antibody titers in ELISA following the vaccination, compared with a placebo | at days 0, 1, 14, 20, 35, 42, 90, 180, 270
  • The proportion of volunteers with increased levels of the immune response in terms of specific neutralizing antibody titers in ELISA greater than ≥ 4 times 21 days following the second vaccination and 90, 180 and 270 days following the first vaccination, compared with a placebo.
The proportion of volunteers with an ex vivo cellular immune response following the vaccination, compared with a placebo | at days 0, 1, 14, 20, 35, 42, 90, 180, 270
  • The proportion of volunteers with an ex vivo cellular immune response 21 days following the second vaccination and 90, 180 and 270 days following the first vaccination, compared with a placebo.
Incidence and type of adverse events during the study | throughout the study, an average of 270 days
  • Immediate adverse events (allergic reactions) that occur within 2 hours after vaccination and that are identified both by the clinical investigator and based on information provided by the volunteer;
  * adverse events (local and systemic reactions) that occur within 7 days after vaccination and that are identified both by the clinical investigator and based on information provided by the volunteer;
  * other adverse events that occur 7 days after each vaccination (from 8 to 42 days after the first vaccination, excluding the allowable interval of visits) and noted by the volunteer in the Self-observation Diary.
Incidence of serious adverse events during the study | throughout the study, an average of 270 days
  • Incidence of serious adverse events during the study.
Cases of early termination of the study due to the development of adverse events / sever adverse events | throughout the study, an average of 270 days
  • Cases of early termination of participation of volunteers in the study due to the development of adverse events / sever adverse events associated with the use of products under study.

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir I. Kuzubov, Principal Investigator — FGBUZ MSCH-163, FMBA of Russia
Locations (1):
- Federal State Budgetary Institution of Healthcare "Medical and Sanitary Unit No. 163 of the Federal Medical and Biological Agency" (FGBUZ MSCH-163, FMBA of Russia), Kol'tsovo, Novosibirsk Oblast, Russia

IPD SHARING:
Plan to Share IPD: No